CLINICAL TRIAL: NCT00653861
Title: Safety and Effectiveness of JUVÉDERM™ Injectable Gel With Lidocaine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allergan Medical (Industry)
Responsible Party: Sponsor
Organization: Allergan (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: JULIDO-001
Record Dates: First submitted 2008-04-02; First posted 2008-04-07 (Estimated); Results first posted 2009-12-30 (Estimated); Last update posted 2014-10-13 (Estimated); Status verified 2013-12

CONDITIONS: Nasolabial Folds
Keywords: Aesthetic correction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Juvederm with Lidocaine (Experimental): Subjects receive Juvederm with Lidocaine (either Ultra or Ultra Plus at investigator's discretion) in one nasolabial fold.
  Interventions: Device: JUVÉDERM™ Injectable Gel with Lidocaine
- Juvederm (Active Comparator): Subjects receive Juvederm without Lidocaine (either Ultra or Ultra Plus at investigator's discretion) in the other nasolabial fold.
  Interventions: Device: JUVÉDERM™ Injectable Gel

INTERVENTIONS:
Device: JUVÉDERM™ Injectable Gel with Lidocaine — Single treatment, volume determined by investigator
  Arms: Juvederm with Lidocaine
Device: JUVÉDERM™ Injectable Gel — Single treatment, volume determined by investigator
  Arms: Juvederm

SUMMARY:
Safety and effectiveness of JUVÉDERM™ Injectable Gel with Lidocaine compared to JUVÉDERM™ without Lidocaine for procedural pain in the treatment of nasolabial folds.

DETAILED DESCRIPTION:
Controlled, randomized, split-face study in which subjects receive JUVÉDERM™ Injectable Gel with Lidocaine (Ultra or Ultra Plus) in one nasolabial fold and JUVÉDERM™ Injectable Gel without Lidocaine (Ultra or Ultra Plus) in the other nasolabial fold. The investigator determines whether the subject receives JUVÉDERM™ Ultra or Ultra Plus per the level of correction desired; the lidocaine assignment is randomized.

ELIGIBILITY:
Inclusion Criteria:

* Be male or female, 18 years of age or older
* Desire correction of moderate to severe nasolabial folds (NLFs)
* Have approximately symmetrical NLFs, i.e., both NLFs have the same pretreatment NLF severity score

Exclusion Criteria:

* Have undergone cosmetic facial procedures in the lower 2/3 of the face within 1 month prior to entry in the study or are planning to undergo these procedure during the study.
* Begin use of any new over-the-counter or prescription, oral or topical, anti-wrinkle products in the NLF area within 1 month prior to enrollment or are planning to begin use of such products during the study.
* Have undergone previous hyaluronic acid (HA)-based dermal filler treatments such that the total volume of HA injected within 12 months prior to study entry is within 5 mL of the recommended annual maximum volume for HA dermal fillers.
* Has ever received semi-permanent fillers or permanent facial implants anywhere in the face or neck, or is planning to be implanted with these products during the study.
* Have a history of anaphylaxis, multiple severe allergies, atopy, or allergy to lidocaine (or any amide-based anesthetic), hyaluronic acid products, or Streptococcal protein, or have plans to undergo desensitization therapy during the term of the study.
* Have an active inflammation, infection, cancerous or pre-cancerous lesion, or unhealed wound in the NLF area

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2008-04; Primary Completion 2008-06 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Mount Kisco, New York, United States

REFERENCES:
- [Result] Weinkle SH, Bank DE, Boyd CM, Gold MH, Thomas JA, Murphy DK. A multi-center, double-blind, randomized controlled study of the safety and effectiveness of Juvederm injectable gel with and without lidocaine. J Cosmet Dermatol. 2009 Sep;8(3):205-10. doi: 10.1111/j.1473-2165.2009.00451.x. PMID 19735519

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Other aesthetic procedures and products were not allowed 1 month prior to study entry or any time during the study.
Groups:
- Total Study Participants: Subjects who received Juvederm with Lidocaine in one nasolabial fold and Juvederm without Lidocaine in the other nasolabial fold
Period: Overall Study
Arm/Group | Total Study Participants
Started | 72
Completed | 72
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Total Study Participants: Subjects who received Juvéderm with Lidocaine in one nasolabial fold and Juvéderm without Lidocaine in the other nasolabial fold.
Arm/Group | Total Study Participants
Number analyzed (Participants) | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 67
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.9 (9.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 72

OUTCOME MEASURES:

1. Primary Outcome: Procedural Pain Score
Description: Evaluate pain on an 11-point scale, where 0 is no pain and 10 is the worst pain imaginable.
Time Frame: 1 day
Population: Intention to treat (ITT)
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Juvéderm Lidocaine Nasolabial Folds (NLFs): Nasolabial folds on one side of the face injected with the Juvederm formulation with lidocaine
- Juvéderm Nasolabial Folds (NLFs): Nasolabial folds on the corresponding side of the face injected with Juvederm
Arm/Group | Juvéderm Lidocaine Nasolabial Folds (NLFs) | Juvéderm Nasolabial Folds (NLFs)
Number analyzed (Participants) | 72 | 72
Units on a scale | 2.0 (1.71) | 5.4 (2.23)

2. Secondary Outcome: Comparative Pain
Description: A 5-point scale (-2 = Right NLF more painful than Left NLF; -1 = Right NLF slightly more painful than Left NLF; 0 = No difference; 1 = Left NLF slightly more painful than Right NLF; 2 = Left NLF more painful than Right NLF). Subjects selected one category from the scale; the percentage of subjects that selected each category is presented.
Time Frame: 1 day
Population: ITT
Measure: Number; unit: Percent of Participants
Arm/Group | Total Study Participants
Number analyzed (Participants) | 72
Percent of Participants
  Juvéderm Lidocaine is Less Painful than Juvéderm | 64
  Juvéderm Lidocaine is Slightly Less Painful | 29
  No Difference | 0
  Juvéderm Lidocaine is Slightly More Painful | 4
  Juvéderm Lidocaine is More Painful than Juvéderm | 3

3. Secondary Outcome: Nasolabial Fold (NLF) Severity
Description: Determination of improvement in NLF severity score on 5-point NLF Severity Scale (0 = None; 1 = Mild; 2 = Moderate; 3 = Severe; 4 = Extreme) two weeks after treatment with Juvederm with Lidocaine (either Ultra or Ultra Plus) in one nasolabial fold and Juvederm (either Ultra or Ultra Plus) in the other nasolabial fold.
Time Frame: 2 weeks
Population: ITT
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Juvéderm Lidocaine NLFs: Nasolabial folds on one side of the face injected with the Juvederm formulation with lidocaine
- Juvéderm NLFs: Nasolabial folds on the corresponding side of the face injected with Juvederm
Arm/Group | Juvéderm Lidocaine NLFs | Juvéderm NLFs
Number analyzed (Participants) | 72 | 72
Units on a scale
  Improvement using Juvederm Ultra | 1.6 (0.60) | 1.6 (0.56)
  Improvement using Juvederm Ultra Plus | 1.8 (0.58) | 1.8 (0.65)

ADVERSE EVENTS:
Arm/Group | Juvéderm Lidocaine Nasolabial Folds (NLFs) | Juvéderm Nasolabial Folds (NLFs)
Serious Adverse Events (participants affected / at risk) | 0/72 | 0/72
Other Adverse Events (participants affected / at risk) | 21/72 | 20/72
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Juvéderm Lidocaine Nasolabial Folds (NLFs) (N=72) | Juvéderm Nasolabial Folds (NLFs) (N=72)
Injection side induration (General disorders) | 11 (11) | 11 (11)
Injection site nodule (General disorders) | 11 (11) | 12 (12)
Injection site discoloration (General disorders) | 8 (8) | 6 (6)
Application site bruising (General disorders) | 6 (6) | 5 (5)
Injection site erythema (General disorders) | 5 (5) | 5 (5)
Injection site edema (General disorders) | 4 (4) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At least ninety (90) days prior to any proposed submission for publication or presentation of Study data or other findings related to the Study, the Investigator will provide the Sponsor with a manuscript of such submission(s) for review and comment.